CLINICAL TRIAL: NCT06707285
Title: MRI Imaging Assessment of Femoral Notch Morphology in Patients With ACL Injury
Brief Title: MRI Morphology of Femoral Notch in ACL Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marian Michel Fahmy Younan, Resident doctor, Assiut University
Other Study IDs: MRI in ACL injury
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: ACL Injury
Keywords: ACL ,femoral notch
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL injured group , non-injured group
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — 1.5T siemens

SUMMARY:
This study aims to investigate the association between femoral notch morphology, as assessed by MRI, and the risk of ACL injury

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18-50 years.
* diagnosed with an ACL injury and confirmed by MRI and age-matched controls.

Exclusion Criteria:

* age <18 yo and >50 years
* patients with previous knee surgeries
* congenital knee deformities
* systemic conditions affecting bone health

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will include adult patients with ACL injury that had previous knee MRI imaging with no history of previous knee surgery or any pathological condition affecting bone health.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between femoral notch morphology and incidence of ACL injury | Base line
  Identify the different types of femoral notch angle , shapes and calculate the notch width index and correlate these differences with the incidence of ACL injury

REFERENCES:
- [Background] Huang M, Li Y, Li H, Liao C, Xu H, Luo X. Predictive effects of the intercondylar notch morphology on anterior cruciate ligament injury in males: A magnetic resonance imaging analysis. Medicine (Baltimore). 2020 Mar;99(10):e19411. doi: 10.1097/MD.0000000000019411. PMID 32150091
- [Background] Micicoi G, Jacquet C, Khakha R, LiArno S, Faizan A, Seil R, Kocaoglu B, Cerciello S, Martz P, Ollivier M. Femoral and Tibial Bony Risk Factors for Anterior Cruciate Ligament Injuries Are Present in More Than 50% of Healthy Individuals. Am J Sports Med. 2021 Dec;49(14):3816-3824. doi: 10.1177/03635465211050421. Epub 2021 Oct 28. PMID 34710345
- [Background] Gultekin MZ, Dincel YM, Keskin Z, Arslan S, Yildirim A. Morphometric risk factors effects on anterior cruciate ligament injury. Jt Dis Relat Surg. 2023;34(1):130-137. doi: 10.52312/jdrs.2023.910. Epub 2022 Dec 27. PMID 36700274
- [Background] Misir A, Sayer G, Uzun E, Guney B, Guney A. Individual and Combined Anatomic Risk Factors for the Development of an Anterior Cruciate Ligament Rupture in Men: A Multiple Factor Analysis Case-Control Study. Am J Sports Med. 2022 Feb;50(2):433-440. doi: 10.1177/03635465211062594. Epub 2022 Jan 12. PMID 35019732
- [Background] Pradhan P, Kaushal SG, Kocher MS, Kiapour AM. Development of Anatomic Risk Factors for ACL Injuries: A Comparison Between ACL-Injured Knees and Matched Controls. Am J Sports Med. 2023 Jul;51(9):2267-2274. doi: 10.1177/03635465231177465. Epub 2023 Jun 13. PMID 37310177
- [Background] Barnum MS, Boyd ED, Vacek P, Slauterbeck JR, Beynnon BD. Association of Geometric Characteristics of Knee Anatomy (Alpha Angle and Intercondylar Notch Type) With Noncontact ACL Injury. Am J Sports Med. 2021 Aug;49(10):2624-2630. doi: 10.1177/03635465211023750. Epub 2021 Jul 8. PMID 34236929